CLINICAL TRIAL: NCT00207051
Title: Phase I Dose Escalation Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of BMS-582664 in Combination With Full Dose Erbitux in Patients With Advanced Gastrointestinal Malignancies Who Have Failed Prior Therapy
Brief Title: BMS-582664 in Combination With Erbitux in Patients With Advanced Gastrointestinal Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA182-003
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-03

CONDITIONS: Colorectal Cancer
Keywords: Advanced Gastrointestinal Malignancies
MeSH Terms: conditions — Colorectal Neoplasms | interventions — brivanib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Brivanib + Cetuximab

INTERVENTIONS:
Drug: Brivanib + Cetuximab — Tablets/IV, Oral/IV , Brivanib 800 mg + Erbitux 400 mg/m2 X 1, followed by 250mg/m2, Brivanib QD / Erbitux QW, up to 48 weeks
  Other Names: Erbitux; BMS-564717

SUMMARY:
This is a phase I dose escalation study to determine the safety, pharmacokinetics and pharmacodynamics of BMS-582664 in combination with full dose erbitux in patients with advanced colorectal cancer who have received no more than 2 prior regimens for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced or metastatic (tumor has spread) gastrointestinal malignancy
* Feeling well other than cancer diagnosis (ie lab work, no infection, etc)
* Available tumor tissue sample from prior surgery
* Measurable disease on scans
* 4-6 weeks since prior therapy and recovered from the effects of prior therapy
* Men and women, ages 18 and above
* Women must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety assessment | throughout the study
dose limiting toxicity (DLT) | assessed for individual patients from C1D1 to C1D28 during the dose escalation portion of the protocol, until maximum tolerated dose is identified
determination of maximum tolerated dose (MTD) | during dose escalation portion of the protocol. Three to six subjects are treated at a specified dose level. If deemed safe dose escalation continues until the maximu tolerated dose is identified

SECONDARY OUTCOMES:
Efficacy based on duration of response and time to progression based on assessment | Measured every 8 weeks throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (5):
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - Georgetn Univ Lombardi Can Ctr, Washington D.C., District of Columbia
  - University Of Miami Miller School Of Medicine, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
- Canada (2):
  - Local Institution, Hamilton, Ontario
  - Local Institution, Toronto, Ontario
- Local Institution, Amsterdam, Netherlands

REFERENCES:
- [Derived] Jonker DJ, Rosen LS, Sawyer MB, de Braud F, Wilding G, Sweeney CJ, Jayson GC, McArthur GA, Rustin G, Goss G, Kantor J, Velasquez L, Syed S, Mokliatchouk O, Feltquate DM, Kollia G, Nuyten DSA, Galbraith S. A phase I study to determine the safety, pharmacokinetics and pharmacodynamics of a dual VEGFR and FGFR inhibitor, brivanib, in patients with advanced or metastatic solid tumors. Ann Oncol. 2011 Jun;22(6):1413-1419. doi: 10.1093/annonc/mdq599. Epub 2010 Dec 3. PMID 21131369
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx